CLINICAL TRIAL: NCT03081858
Title: A Phase 1/2a Pilot Study of Intravesical TSD-001 for Treatment of Low-Grade, Stage Ta, Non Muscle Invasive Bladder Cancer
Brief Title: Proliposomal Intravesical Paclitaxel for Treatment of Low-Grade, Stage Ta, Non Muscle Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lipac Oncology LLC (Industry)
Collaborators: TesoRx Pharma, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TD-001
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Bladder Cancer Cell Transitional; Non-Muscle Invasive Bladder Cancer; Bladder Cancer; Urinary Bladder; Transitional Cell Carcinoma of the Bladder; Urinary Bladder Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Urinary Bladder Diseases; Urologic Diseases
Keywords: NMIBC; Paclitaxel; Antineoplastic Agents; Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Urinary Bladder Diseases; Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TSD-001 Administration Part 1, Cohort 1 (Experimental): Part 1, Cohort 1: For the first 3 subjects enrolled, the initial dose will be 10 mg in Sterile Water for Injection (SWFI). TSD-001 will be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on subject's tolerability of the procedure). If Dose Limiting Toxicity(DLT) does not develop, intravesical instillation 14 days later will be titrated up according to the schedule (25, 50, 75, 100, 150 mg in SWFI) until DLT (defined as any grade 3 or 4 toxicity or prolonged [greater than 14 days] grade 2 toxicity) is observed.
  Interventions: Drug: TSD-001
- TSD-001 Administration Part 1, Cohort 2 (Experimental): Part 1, Cohort 1: For the next 3 subjects enrolled, the initial dose will be 90 mg in SWFI. TSD-001 will be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on subject's tolerability of the procedure). If DLT does not develop, intravesical instillation 14 days later will be titrated up according to the schedule (180, 270, 360, 450, and 540 mg in SWFI) until DLT (defined as any grade 3 or 4 toxicity or prolonged [greater than 14 days] grade 2 toxicity) is observed.
  If no DLT is observed in the first 6 subjects (cohorts 1 and 2) after titration up to 540 mg, then the maximum deliverable dose (MDD) will be defined and dose recommended for part 2 of the study.
  Interventions: Drug: TSD-001
- TSD-001 Administration Part 2 (Experimental): In part 2, the dose will be selected as the MTD/MDD, established in part 1 and provided weekly via the intravesical route.
  During part 2, up to 10 additional subjects will receive intravesical instillations of TSD-001 via urethral catheterization of the urinary bladder at the MTD/MDD established in part 1 at weekly intervals for 6 consecutive weeks. TSD-001 will be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on subject's tolerability of the procedure).
  Interventions: Drug: TSD-001

INTERVENTIONS:
Drug: TSD-001 — Administered via intravesical instillation.
  Other Names: Proliposomal Intravesical Paclitaxel

SUMMARY:
This is a single-arm, phase 1/2a study of formulated paclitaxel in subjects with low-grade, noninvasive papillary carcinoma (stage Ta) of the bladder.

Part 1 of the study will enroll 6 subjects (3 per cohort) with low-grade, stage Ta transitional cell carcinoma (TCC) of the bladder who will receive escalating doses of paclitaxel formulated as TSD-001 every 2 weeks for 6 treatments until Dose Limiting Toxicity (or until the Maximum Deliverable Dose) is observed (Maximum Tolerated Dose established).

Part 2 of the study will enroll an additional 10 subjects with low-grade, stage Ta (uni-or multifocal) TCC of the bladder who will receive weekly TSD-001 for 6 weeks at the highest nontoxic dose (i.e., MTD) established in part 1 of the study. May meet definition of low grade without histological tissue diagnosis if on cystoscopic assessment they have a solitary papillary tumor.

Part 3 of the study will continue to track subjects enrolled in Parts 1 and 2 to determine rates of disease-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of low grade (G1 or G2), uni- or multifocal papillary appearing bladder tumor, stage Ta.
* For part 1, subject will have ≥ 1 and ≤ 5 tumors (prior to TURBT), none of which exceeds 3.0 cm in diameter; for part 2, patient will have ≥ 2 and ≤ 5 tumors (prior to TURBT), none of which exceeds 3.0 cm in diameter (resection loop ~1 cm), OR, for part 2, subject meets this inclusion if on cystoscopic assessment they have a solitary papillary tumor (> 0.5 cm and ≤ 2.0 cm in diameter)..
* Subject is surgical candidate for TURBT as part of normal NMIBC treatment plan. For part 1, successful completion of TURBT procedure. For part 2, successful completion of cystoscopic assessment/TURBT procedure with one marker lesion left intact; the marker lesion should be > 0.5 cm and < 2.0 cm in diameter.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Peripheral neuropathy grade 1 or less.
* Adequate hematological, hepatic, and renal parameters; i.e., hemoglobin > 10 g/dL, creatinine < 3.5 mg/dL, bilirubin < 1.5 mg/dL , and aspartate aminotransferase, alanine aminotransferase < 50 U/L, and alkaline phosphatase < 130 U/L.
* All sexually active subjects of reproductive potential are required to use or start using a reliable method of birth control at least 2 weeks prior to study enrollment, throughout the study, and for at least 3 months following completion of study therapy.
* Females of childbearing potential must have a negative pregnancy test within 30 days prior to enrollment. Females who are postmenopausal for at least 1 year (defined as more than 12 months since last menses) or are surgically sterilized do not require this test.
* For male subjects, the digital rectal examination must not be suspicious for carcinoma of the prostate.
* Able to retain bladder instillations for up to 120 minutes (± 15 minutes).

Exclusion Criteria:

* Has an active concurrent malignancy/life-threatening disease. If there is a history of prior malignancies/life-threatening diseases, the subject is to be disease free for at least 5 years. Subjects with other prior malignancies less than 5 years before study entry may still be enrolled if they have received treatment resulting in complete resolution of the cancer and currently have no clinical, radiologic, or laboratory evidence of active or recurrent disease. Subjects will not be excluded for recurrent NMIBC, basal or squamous cell skin cancers, or noninvasive cancer of the cervix.
* Has positive urine cytology for urothelial malignancy at screening.
* Has an active uncontrolled infection, including a urinary tract infection, underlying medical condition, or other serious illness that would impair the ability of the subject to receive protocol treatment.
* Previous intravesical therapy within 6 months of study entry.
* Prior radiation to the pelvis.
* Participated in a previous clinical trial or used any investigational drugs, biologics, or devices within 90 days prior to study treatment or plans to use any of these during the course of the study.
* Has had any previous exposure to paclitaxel or docetaxel in the last 5 years.
* Has or has ever had: upper tract TCC; urethral tumor (prostatic urethra included); any invasive bladder tumor known to be other than tumor Ta, low-grade (G1-G2); any evidence of lymph node or distant metastasis; any bladder tumor with histology other than TCC; or carcinoma in situ (CIS).
* Has a tumor in a bladder diverticulum
* Concurrent treatment with any chemotherapeutic agent.
* History of vesicoureteral reflux.
* An indwelling ureteral stent.
* Has received any pelvic radiotherapy (including external beam and/or brachytherapy.)
* Has a bleeding disorder or a screening platelet count < 100×109/L.
* Has an active diagnosis of interstitial cystitis.
* For subjects with recurrent tumor, the subject had at least a 6-month cystoscopically confirmed tumor-free interval between the last tumor recurrence and screening cystoscopic examination.
* Presence of poorly controlled diabetes mellitus (glycated hemoglobin [HgbA1c] > 9.0%).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2021-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Oefelein, MD, Study Director — Lipac Oncology LLC
Locations (5):
- United States (5):
  - Urological Associates of Southern Arizona, PC, Tucson, Arizona
  - Trovare Clinical Research, Bakersfield, California
  - Tower Urology, Los Angeles, California
  - Chesapeake Urology Associates, Hanover, Maryland
  - Carolina Urologic Research Clinic, Myrtle Beach, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TSD-001 Administration Part 1, Cohort 1: Part 1, Cohort 1: For the first 3 subjects enrolled, the initial dose was 10 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure). As Dose Limiting Toxicity(DLT) did not develop, intravesical instillation 14 days later was titrated up according to the schedule (25, 50, 75, 100, 150 mg in SWFI).
  TSD-001: Administered via intravesical instillation.
- TSD-001 Administration Part 1, Cohort 2: Part 1, Cohort 2: For the next 3 subjects enrolled, the initial dose was 90 mg in SWFI. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure). As DLT did not develop, intravesical instillation 14 days later was titrated up according to the schedule (180, 270, 360, 450, and 540 mg in SWFI).
  As no DLT was observed in the first 6 subjects (cohorts 1 and 2) after titration up, the maximum deliverable dose (MDD) was defined as 360 mg and the dose was recommended for part 2 of the study.
  TSD-001: Administered via intravesical instillation.
- TSD-001 Administration Part 2, Cohort 1: In part 2, cohort 1, the dose administered was planned as the MDD established in part 1, and provided weekly via the intravesical route.
  During part 2, cohort 1, 6 additional subjects received intravesical instillations of TSD-001 via urethral catheterization of the urinary bladder at the MDD established in part 1 at weekly intervals for 6 consecutive weeks. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure).
  TSD-001: Administered via intravesical instillation.
- TSD-001 Administration Part 2, Cohort 2: In part 2, cohort 2, the dose was selected as the MDD, established in part 1, and provided weekly via the intravesical route.
  During part 2, cohort 2, 3 additional subjects received intravesical instillations of TSD-001 via urethral catheterization of the urinary bladder at the MDD established in part 1 at weekly intervals for 8 consecutive weeks. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure).
  TSD-001: Administered via intravesical instillation.
Period: Overall Study
Arm/Group | TSD-001 Administration Part 1, Cohort 1 | TSD-001 Administration Part 1, Cohort 2 | TSD-001 Administration Part 2, Cohort 1 | TSD-001 Administration Part 2, Cohort 2
Started | 3 | 3 | 6 | 3
Completed | 1 | 3 | 6 | 3
Not Completed | 2 | 0 | 0 | 0
Not completed — Sponsor Discontinuation - IP issue for investigation (Bacterial Endotoxin level) | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TSD-001 Administration Part 2, Cohort 1: In part 2, cohort 1, the MDD of 360 mg, established in part 1, was provided weekly via the intravesical route.
  During part 2, cohort 1, 6 additional subjects received intravesical instillations of TSD-001 via urethral catheterization of the urinary bladder at the MDD established in part 1 at weekly intervals for 6 consecutive weeks. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure).
  TSD-001: Administered via intravesical instillation.
- TSD Administration Part 2, Cohort 2: In part 2, cohort 1, the MDD of 360 mg, established in part 1, was provided weekly via the intravesical route.
  During part 2, cohort 2, 3 additional subjects received intravesical instillations of TSD-001 via urethral catheterization of the urinary bladder at the MDD established in part 1 at weekly intervals for 8 consecutive weeks. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure).
  TSD-001: Administered via intravesical instillation.
- Total: Total of all reporting groups
Arm/Group | TSD-001 Administration Part 1, Cohort 1 | TSD-001 Administration Part 1, Cohort 2 | TSD-001 Administration Part 2, Cohort 1 | TSD Administration Part 2, Cohort 2 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.33 (8.96) | 71.67 (5.51) | 57.50 (16.99) | 64.33 (17.79) | 65.27 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 4 | 0 | 5
  Male | 3 | 2 | 2 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White/ Not Hispanic or Latino | 3 | 2 | 4 | 3 | 12
  Race/Ethnicity: Asian/ Not Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Race/Ethnicity: White/ Hispanic or Latino | 0 | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 3 | 15
Non-Muscle Invasive Bladder Cancer Recurrent [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 6 | 3 | 12
  No | 2 | 1 | 0 | 0 | 3
Number of Tumor Locations [Count of Participants; unit: Participants]
  Solitary | 2 | 1 | 2 | 0 | 5
  Multifocal | 1 | 2 | 4 | 3 | 10
Previous Intravesical Therapy [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 3 | 2 | 6
  No | 2 | 3 | 3 | 1 | 9
European Association of Urology (EAU) Risk Stratification [Count of Participants; unit: Participants] — Low risk defined as: Primary, Solitary, low-grade (LG)/grade 1 (G1)<3cm, no carcinoma in situ (CIS)
  Intermediate risk defined as: All tumors not defined in the two adjacent categories
  High risk defined as any of the following:
  * T1 stage tumor
  * high-grade/grade 3 (HG/G3) tumor
  * CIS
  * Multiple, recurrent, and large (>3cm) Ta tumor/low-grade (grade 1/Grade 2) (Ta G1/G2) tumors (all conditions present)
  Participants
    Low Risk | 2 | 0 | 0 | 0 | 2
    Intermediate Risk | 1 | 3 | 6 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Tolerated Dose or Maximum Deliverable Dose (MDD)
Description: Dose immediately preceding the dose at which DLT occurs or when a MDD is reached.
Time Frame: 12 weeks
Population: MITT/PK Population
Measure: Number; unit: mg
Arm/Group | TSD-001 Administration Part 1, Cohort 1 | TSD-001 Administration Part 1, Cohort 2
Number analyzed (Participants) | 3 | 3
mg | NA — MTD and/or MDD was not reached in dose escalation in Part 1, Cohort 1 patient treatments. | 360

2. Primary Outcome: Part 2: Marker Lesion Response Rate
Description: Determine the marker lesion response rate at final assessment visit for subjects that received the MDD established in part 1.
Time Frame: 12 weeks (Cohort 1) or 15 weeks (Cohort 2)
Population: Per Protocol (PP) Population: The PP population will include subjects in the MITT population who have no major protocol violations.
  Note: Modified Intent-to-Treat (MITT) population includes all enrolled subjects who received at least one dose of study drug and have at least one post-baseline measurement of paclitaxel concentration.
Measure: Count of Participants; unit: Participants
Groups:
- TSD-001 Administration Part 2, Cohort 1: In part 2, cohort 1, the MDD of 360 mg was provided weekly via the intravesical route at weekly intervals for 6 consecutive weeks. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more was acceptable, depending on the subject's tolerability of the procedure). Marker lesion response was determined at 12 weeks (± 7 days) after Day 1.
- TSD Administration Part 2, Cohort 2: In part 2, cohort 2, the MDD of 360 mg, established in part 1, was provided weekly via the intravesical route.
  These subjects received intravesical instillations of TSD-001 via urethral catheterization of the urinary bladder at the MDD established in part 1 at weekly intervals for 8 consecutive weeks. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure). Marker lesion response was determined 15 weeks (± 7 days) after Day 1.
Arm/Group | TSD-001 Administration Part 2, Cohort 1 | TSD Administration Part 2, Cohort 2
Number analyzed (Participants) | 5 | 3
Participants
  Complete Response | 0 | 1
  Partial Response | 3 | 1
  Marker Lesion Response | 3 | 2

3. Secondary Outcome: Part 1: Determine Paclitaxel Concentrations
Description: Determine the local (bladder urine) and systemic (peripheral blood) paclitaxel concentrations before and after intravesical exposure to TSD-001 at all doses. Blood and urine samples were collected 15 (± 15) minutes before and 2 hours (± 10 minutes) after each instillation. Results are presented for different dose levels administered during dose escalation. The remaining results are grouped by cohort.
Time Frame: 10 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/L
Groups:
- TSD-001 Administration Part 1, Cohort 1: Day 1: 10 mg: For these subjects, the initial dose was 10 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 1: Week 2: 25 mg: For these subjects, the second dose was 25 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 1: Week 4: 50 mg: For these subjects, the third dose was 50 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 1: Week 6: 75 mg: For these subjects, the fourth dose was 75 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 1: Week 8: 100 mg: For these subjects, the fifth dose was 100 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 1: Week 10: 150 mg: For these subjects, the sixth dose was 150 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 2: Day 1: 90 mg: For these subjects, the initial dose was 90 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 2: Week 2: 180 mg: For these subjects, the second dose was 180 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 2: Week 4: 270 mg: For these subjects, the third dose was 270 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 2: Week 6: 360 mg: For these subjects, the fourth dose was 360 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 2: Week 8: 450 mg: For these subjects, the fifth dose was 450 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
- TSD-001 Administration Part 1, Cohort 2: Week 10: 540 mg: For these subjects, the sixth dose was 540 mg in Sterile Water for Injection (SWFI). TSD-001 was planned to be retained in the bladder for 1 hour or more (up to 2 hours) as acceptable, depending on the subject's tolerability of the procedure.
Arm/Group | TSD-001 Administration Part 1, Cohort 1: Day 1: 10 mg | TSD-001 Administration Part 1, Cohort 1: Week 2: 25 mg | TSD-001 Administration Part 1, Cohort 1: Week 4: 50 mg | TSD-001 Administration Part 1, Cohort 1: Week 6: 75 mg | TSD-001 Administration Part 1, Cohort 1: Week 8: 100 mg | TSD-001 Administration Part 1, Cohort 1: Week 10: 150 mg | TSD-001 Administration Part 1, Cohort 2: Day 1: 90 mg | TSD-001 Administration Part 1, Cohort 2: Week 2: 180 mg | TSD-001 Administration Part 1, Cohort 2: Week 4: 270 mg | TSD-001 Administration Part 1, Cohort 2: Week 6: 360 mg | TSD-001 Administration Part 1, Cohort 2: Week 8: 450 mg | TSD-001 Administration Part 1, Cohort 2: Week 10: 540 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 1 | 3 | 3 | 3 | 3 | 3 | 3
ug/L
  Predose Urine - Paclitaxel Concentration in Urine collected 15 minutes before | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0) | .8 (1.4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Postdose Urine - Paclitaxel Concentration in Urine collected 2 hrs post: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3
  Postdose Urine - Paclitaxel Concentration in Urine collected 2 hrs post | 19367 (4341) | 72933 (50497) | 189667 (73433) | 287333 (134016) | 436000 | 446000 | 241000 (35539) | 699000 (272567) | 686667 (167861) | 1161667 (760795) | 1800000 (606300) | 1886333 (1317354)
  Predose Plasma - Paclitaxel Concentration in Plasma collected 15 minutes before: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3
  Predose Plasma - Paclitaxel Concentration in Plasma collected 15 minutes before | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Postdose Plasma - Paclitaxel Concentration in Plasma collected 2 hrs post: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1 | 1 | 3 | 3 | 3 | 3 | 3 | 3
  Postdose Plasma - Paclitaxel Concentration in Plasma collected 2 hrs post | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

4. Secondary Outcome: Part 2: Determine Paclitaxel Concentrations
Description: Determine the systemic (peripheral blood) paclitaxel concentrations 15 (± 15) minutes before, and 2 hours (± 10 minutes) after the third intravesical instillation (Week 2) of TSD-001.
Time Frame: Week 2 (pre and post dose)
Population: Per Protocol (PP): This population will include subjects in the MITT population who have no major protocol violations.
  Note: The Modified Intent to Treat (MITT) population includes enrolled subjects who received at least one dose of study drug and have at least one post-baseline measurement of paclitaxel concentration.
Measure: Mean (Standard Deviation); unit: ug/L
Groups:
- TSD-001 Administration Part 2, Cohort 1: In part 2, cohort 1, the MDD of 360 mg was instilled intravesically. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more was acceptable, depending on the subject's tolerability of the procedure).
- TSD-001 Administration Part 2, Cohort 2: In part 2, cohort 2, the MDD of 360 mg was instilled intravesically. TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more was acceptable, depending on the subject's tolerability of the procedure).
Arm/Group | TSD-001 Administration Part 2, Cohort 1 | TSD-001 Administration Part 2, Cohort 2
Number analyzed (Participants) | 5 | 3
ug/L
  Predose | 0 (0) | 0 (0)
  Postdose | 0 (0) | 0 (0)

5. Other Pre Specified Outcome: Part 3: Rates of Recurrence/Disease-Free Survival in Part 1 Subjects Only at 12 and 24 Months
Description: Long-term follow-up to determine when histological tissue diagnosis evidence of recurrence occurs for subjects after complete TURBT and exposure to TSD-001 in part 1. Cystoscopic surveillance was performed every 3 months from the last endoscopic assessment in part 1 until 24 months (from initial TURBT and instillation). Part 2 subjects, different than part 1 subjects, were followed for marker lesion response and did not have standardized TURBT timing to use as a baseline and so are not included in these reported RFS rates.
  Recurrence-free survival is no histological evidence of transitional cell carcinoma (TCC) recurrence in the time outlined for the TCC risk level.
Time Frame: 2 years
Population: The MITT population will include all enrolled subjects who received at least one dose of study drug and had at least one post-baseline measurement of paclitaxel concentration.
Measure: Count of Participants; unit: Participants
Groups:
- TSD-001 Administration Part 1, Cohort 1: Long-term Follow-up (Part 3); TSD-001 Administration Part 1, Cohort 2: Long-term Follow-up (Part 3): Part 1 patients were followed for recurrence free survival (RFS) for up to 2 years after initial TURBT and intravesical exposure to TSD-001. The tracking and recording of RFS occurred in TD-001 part 3, the observational study of recurrence in these patients. Patients enrolled in part 3 underwent standard of care cystoscopy bladder tumor follow-up every 3 months.
Arm/Group | TSD-001 Administration Part 1, Cohort 1: Long-term Follow-up (Part 3) | TSD-001 Administration Part 1, Cohort 2: Long-term Follow-up (Part 3)
Number analyzed (Participants) | 3 | 3
Participants
  One Year: Disease-Free | 3 | 2
  One Year: Recurrence Occurred | 0 | 1
  Two Year: Disease-Free | 3 | 2
  Two Year: Recurrence Occurred | 0 | 1

ADVERSE EVENTS:
Time Frame: For Part 1 patients, the time period for adverse event collection was 16 weeks after the first treatment. For Part 2 patients, the time period for adverse event collection was 13 Weeks after the first treatment. During part 3, AEs continued from part 1 or part 2 will be followed until resolution, stabilization, or end of study, but no new AEs will be recorded (excepts SAEs). So, the total time frame was 2 years from the first treatment.
Description: The severity and frequency of AEs were assessed following administration and defined per the NCI CTCAE Version 5.0. The study was not designed or powered to support formal comparisons of AEs across individual dose levels, so the Statistical Analysis Plan pre-specified the reporting of AEs grouped by each cohort within part 1 and part 2. The continued tracking of AEs and recording of new/continuing SAEs is pre-specified to be for all participants in Part 3 as outlined above.
Groups:
- TSD-001 Administration Part 1, Cohort 1; TSD-001 Administration Part 1, Cohort 2: In part 1, these subjects were treated in a planned six-dose escalation of TSD-001 every 2 weeks via the intravesical route until DLT (establishing MTD) or until MDD was reached.
  TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more was acceptable, depending on the subject's tolerability of the procedure).
- TSD-001 Administration Part 2, Cohort 1: In part 2, cohort 1, the dose administered was planned as the MDD established in part 1, and provided weekly via the intravesical route for six doses.
  TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure).
- TSD-001 Administration Part 2, Cohort 2: In part 2, cohort 2, the dose administered was planned as the MDD established in part 1, and provided weekly via the intravesical route for eight doses.
  TSD-001 was planned to be retained in the bladder for 2 hours (1 hour or more will be acceptable, depending on the subject's tolerability of the procedure).
- TD-001 Part 3 (Long-term Surveillance): All subjects in part 1 and part 2, were eligible for continued surveillance for safety event for up to 2 years after initial intravesical exposure to TSD-001. This observational study of safety (all subjects) and recurrence (Part 1 subjects only) followed standard of care cystoscopy bladder tumor follow-up every 3 months. During this time, only SAEs and those AEs related to SAEs were tracked and recorded.
Arm/Group | TSD-001 Administration Part 1, Cohort 1 | TSD-001 Administration Part 1, Cohort 2 | TSD-001 Administration Part 2, Cohort 1 | TSD-001 Administration Part 2, Cohort 2 | TD-001 Part 3 (Long-term Surveillance)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/6 | 1/3 | 1/10
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 6/6 | 2/3 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSD-001 Administration Part 1, Cohort 1 (N=3) | TSD-001 Administration Part 1, Cohort 2 (N=3) | TSD-001 Administration Part 2, Cohort 1 (N=6) | TSD-001 Administration Part 2, Cohort 2 (N=3) | TD-001 Part 3 (Long-term Surveillance) (N=10)
acute pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Initially presented with a urinary tract infection (UTI) from a multi-resistant E. Coli which failed antimicrobial therapy. The investigator concluded it was not related to study drug, but it was related to study procedure (i.e. catheterization).
Extraperitoneal Bladder abscess (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — In Part 3, follow-up from part 1, patient with recurrent TaN0M0 bladder cancer (intermediate risk category) who was hospitalized for extraperitoneal bladder rupture and abscess due to complications of TURBT. Assessed as severe, unrelated to IP.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TSD-001 Administration Part 1, Cohort 1 (N=3) | TSD-001 Administration Part 1, Cohort 2 (N=3) | TSD-001 Administration Part 2, Cohort 1 (N=6) | TSD-001 Administration Part 2, Cohort 2 (N=3) | TD-001 Part 3 (Long-term Surveillance) (N=10)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 4 (4) | 0 | 0
Fatigue (General disorders) | 0 | 1 (1) | 3 (4) | 1 (1) | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 (3) | 0 | 0
Urinary tract infection (Infections and infestations) | 1 (2) | 0 | 3 (4) | 1 (1) | 0
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 1 (1) | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (3) | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 (2) | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 (1) | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0
Anorgasmia (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 (1) | 1 (1) | 0 | 0
Bladder discomfort (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 (1) | 0 | 0
Extraperitoneal Bladder Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) — Abscess
Abdominal Pain (Infections and infestations) | 0 | 0 | 0 | 0 | 1 (1) — Abdominal Pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least 90 days before the proposed submission for publication/presentation of Study data or findings, the PI will provide the Sponsor with a manuscript for review. No release of confidential information without the Sponsor's written approval. Multi-center results to be published conjointly under Sponsor's direction, but if this final manuscript has not been published within 12 months after study end at all sites, the PI may publish results, subject to contract confidentiality.

DOCUMENTS (2):
  • Study Protocol (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/58/NCT03081858/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT03081858/SAP_001.pdf